CLINICAL TRIAL: NCT00533299
Title: Randomized, Double-Blind, Phase III Trial of Chemotherapy Plus the Transcriptional Therapy Hydralazine and Magnesium Valproate Versus Chemotherapy Plus Placebo in Cisplatin-Resistant Recurrent Ovarian Cancer.
Brief Title: Hydralazine Valproate for Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 006/028/DDI
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2007-09-21 (Estimated); Status verified 2007-08

CONDITIONS: Ovarian Cancer
Keywords: Epigenetics, hydralazine, valproate, ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hydralazine; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Topotecan hydralazine valproate
  Interventions: Drug: Hydralazine and magnesium valproate
- 2 (Placebo Comparator): Placebo, hydralazine, valproate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydralazine and magnesium valproate — Hydralazine and valproate will start from seven days before day 1 of chemotherapy until the end of the sixth course. Hydralazine will be administered at 182mg (rapid) or 83mg (slow) according to the acetylator phenotype in a single daily dose and magnesium valproate at an oral dose of 40mg/Kg t.i.d.
  Arms: 1
Drug: Placebo — Placebos will start from seven days before day 1 of chemotherapy until the end of the sixth course. Placebo tablets will be administered in an identical form that experimental drugs.
  Arms: 2

SUMMARY:
The current standard for recurrent, persistent or metastatic cisplatin-resistant ovarian cancer is palliative chemotherapy with either topotecan, liposomal doxorubicin or gemcitabine, however, the results need to be improved. Epigenetic aberrations play an important role in cancer progression by silencing growth regulatory genes and there is now evidence that inhibitors of DNA methylation and HDAC inhibition synergize the cytotoxicity of chemotherapy.

Objective. To determine the superiority of epigenetic therapy with hydralazine and valproate plus topotecan over placebo plus topotecan upon progression-free survival.

Hypothesis. Hydralazine and magnesium valproate associated to topotecan will increase progression-free survival from 6 to 9 months as compared with the same regimen of chemotherapy plus placebo.

DETAILED DESCRIPTION:
Randomized, double-blind phase III trial. A total of 211 patients (alpha 0.5, power 0.8)with cisplatin-resistant recurrent or persistent cancer will be randomized to topotecan + placebo or topotecan + hydralazine + valproate for 6 courses every 4 weeks. Patients will receive an oral dose of hydralazine of 182mg (rapid) or 83mg (slow) according to the acetylator phenotype in a single daily dose and magnesium valproate at an oral dose of 40mg/Kg t.i.d. Both drugs in a slow-release formulation. Experimental drugs or placebo will start from seven days before day 1 of chemotherapy until the end of the sixth course.

ELIGIBILITY:
Inclusion Criteria:

* Measurable or evaluable disease(evaluable according to CA125 criteria of GCIG) Cisplatin resistant ovarian cancer
* Persistent or progression to first line platinum-based chemotherapy
* Relapse within 6 months after completing first line platinum-based chemotherapy
* Platinum-sensitive disease who are failed to second line therapy based on platinum.
* Adequate organic function as defined by: hemoglobin >10 g/L, leukocytes >4000/mm3, platelets >100 000mm3; normal creatinine value and creatinine clearance >60 mL/min; total bilirubin < 1.5 upper normal limit value

Exclusion Criteria:

* History of allergy to hydralazine or valproate;
* Past or present condition of rheumatic disease, central nervous system disease, heart failure from aortic stenosis and postural hypotension as diagnosed by a physician;
* Newly diagnosed hypertension patients with or without pharmacological treatment are allowed as long as their treatment do not include hydralazine.
* Previous use of the experimental drugs (hydralazine and magnesium valproate) as well as if patients were pregnant or breast-feeding.

Other exclusion criteria are uncontrolled systemic disease or infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2007-08; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 2-years

SECONDARY OUTCOMES:
Safety, response, overall survival. | 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Gallardo, MD, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Tlalpan, Mexico